CLINICAL TRIAL: NCT00154765
Title: Graduate School of Physical Therapy, College of Medicine, NTU, Taiwan
Brief Title: Effect of Sling Suspension Exercises in Proprioception of Patients With Knee Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Educational/Counseling/Training
Other Study IDs: 9100207243
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Last update posted 2005-11-22 (Estimated); Status verified 2003-12

CONDITIONS: Osteoarthritis
MeSH Terms: conditions — Osteoarthritis

INTERVENTIONS:
Device: sling suspension exercises

SUMMARY:
Therapeutic exercise is important to patients with knee osteoarthritis. Few studies reported the effect of therapeutic exercise in proprioception for these patients. The purposes of this study were to investigate the training effect of sling suspension exercises, as a proprioception-training tool, for patients with knee osteoarthritis and further, to build up an model of proprioception training.

DETAILED DESCRIPTION:
Therapeutic exercise is important to patients with knee osteoarthritis. Few studies reported the effect of therapeutic exercise in proprioception for these patients. The purposes of this study were to investigate the train-ing effect of sling suspension exercises, as a proprioception-training tool, for patients with knee osteoarthritis and further, to build up an model of proprioception training. Twelve subjects were recruited in this study. The inclusion criteria were aged 50 to 70, both genders, diagnosed as knee osteoarthritis, grading 2 or 3 in Kellgren's scale. After having their consents all subjects received baseline measurements including active joint reposition test, functional ambulating test and self-evaluating with Western Ontario & McMaster Universities Arthritis Index (WOMAC). Then they were randomly assigned to training group and reference group. Seven subjects in the training group received the treatment of heat, interferential current (IFC), and sling suspension exercises or just only sling suspension exercises. Five subjects in the reference group received the treatment of heat and IFC or no intervention. The training sessions of sling suspension exercises were 3 times per week, lasting for8 weeks. After 8-week training, both groups were given post-test which is completely the same as pre-test. Mann-Whitney U Test was used to test the difference between groups, and Wilcoxon Signed Ranks Test was used to test pre-post difference in both groups. The results showed it was no difference between both groups in all the measurements of pre-test. After 8 weeks, it showed significant difference on joint reposi-tion test (p<.05) but no difference on functional ambulating test and WOMAC index (p>.05) between the 2 groups. In the training group, all mea-surements got significant improvement (p<.05) except one of the functional ambulating tests. However, the reference group only showed significant improvement in pain and physical function subscales of WOMAC (p<.05). This study concludes that the sling suspension exercises designed for patients with knee osteoarthritis improve the proprioception of knee joint. The con-tent and concept of sling suspension exercises in this study might be a refer-ence of proprioception training for patients with knee osteoarthritis. Increasing case number and elongating the duration of intervention are suggested in further studies.

ELIGIBILITY:
Inclusion Criteria:

* aged 50 to 70, both genders, diagnosed as knee osteoarthritis, grading 2 or 3 in Kellgren's scale

Exclusion Criteria:

-

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30
Dates: Start 2003-03; Study Completion 2003-12

PRIMARY OUTCOMES:
Significant difference on joint reposi-tion test (p<.05)
No difference on functional ambulating test and WOMAC index (p>.05) between the 2 groups.
In the training group, all mea-surements got significant improvement (p<.05) except one of the functional ambulating tests.

CONTACTS AND LOCATIONS:
Overall Officials: J Y Tsauo, PhD, Study Director — Grad School of PT, Collegeof Medicine, NTU
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan